CLINICAL TRIAL: NCT07075393
Title: Description of Renal Involvement in Wilson's Disease
Acronym: WILKID
Status: Not yet recruiting | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: APS_2025_1
Record Dates: First submitted 2025-07-11; First posted 2025-07-20 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Wilson Disease
MeSH Terms: conditions — Hepatolenticular Degeneration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Wilson disease patients: Patients followed for wilson disease
  Interventions: Other: full renal workup

INTERVENTIONS:
Other: full renal workup — full renal workup (biology and echography)

SUMMARY:
Wilson's disease (WD) is a rare genetic disorder that leads to copper accumulation in various tissues, including the liver, nervous system, heart, and kidneys. Renal involvement in WD has been poorly studied, and systematic screening is not currently recommended.

Indirect renal complications are the most common, such as hepatorenal and cardiorenal syndromes, as well as severe complications like hemolysis or rhabdomyolysis. However, literature suggests that copper may exert a direct toxic effect on renal tubular cells, leading to both proximal and distal tubular dysfunction. These may manifest through often subtle signs, such as aminoaciduria, glycosuria, hypouricemia, and low-molecular-weight proteinuria. Electrolyte imbalances of varying severity may also occur, including hypokalemia, which can cause muscle cramps and cardiac arrhythmias, as well as acid-base disorders (proximal or distal renal tubular acidosis), and/or phosphate-calcium metabolism abnormalities (phosphate diabetes and hypercalciuria). These latter issues may lead to complications such as urinary stones, nephrocalcinosis, and even fracture-related osteoporosis.

In addition, long-term treatment with D-penicillamine (DPA), a common therapy for WD, can cause renal damage in 10-20% of cases, mainly affecting the glomeruli. This includes membranous nephropathy, severe proliferative glomerulonephritis, or nephrotic syndrome with minimal change disease.

Without appropriate monitoring and preventive care, both direct and indirect renal complications can lead to acute or chronic kidney failure. It is likely that the prevalence and systemic impact of renal involvement in WD are currently underestimated.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 7 years and older
* Diagnosed with Wilson's disease, with a Leipzig score ≥ 4

Exclusion Criteria:

* Patient who has undergone organ transplantation
* Known renal comorbidity unrelated to Wilson's disease
* Pregnant or breastfeeding woman

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients followed for Wilson disease accepting to undergo full renal workup (biology and echography)
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Prevalence of renal involvement in Wilson's disease | Day 0
  Renal involvement is defined by the presence of at least one of the following criteria:
  * Chronic kidney disease, defined by an estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m² and/or proteinuria > 0.5 g/g of creatinine.
  * Markers of proximal tubulopathy, defined by at least one of the following: phosphate diabetes (renal phosphate wasting), hypokalemia, normoglycemic glycosuria, β2-microglobulinuria, hypouricemia, or metabolic acidosis.
  * Hypercalciuria and/or urolithiasis.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Fondation Adolphe de Rothschild, Paris, France